CLINICAL TRIAL: NCT02434393
Title: Characterizing Cognitive Decline in Late Life Depression: The Alzheimer's Disease Neuroimaging Initiative - Depression Project
Brief Title: Characterizing Cognitive Decline in Late Life Depression: The ADNI Depression Project
Acronym: ADNI-D
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Francisco (Other); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Other Study IDs: ADC-048; R01MH098062 (NIH)
Record Dates: First submitted 2014-12-24; First posted 2015-05-05 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Major Depression; Late Life Depression (LLD)
Keywords: Depression; Late Life Depression; LLD; amyloid imaging; biomarkers
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Late Life Depression: 120 participants who meet the criteria for Major Depression or Late Life Depression (LLD)

SUMMARY:
The purpose of this research study is to characterize the mechanisms contributing to cognitive impairment and accelerated cognitive decline in Late Life Depression (LLD).

This is a non-randomized, observational, non-treatment study that originally launched in 2015, enrolling 133 participants. From the originally enrolled participants, the continuation of the ADNI-D study will enroll 120 participants which will include following participants from the original (parent) protocol and enrollment of new participants for a period of 30 months. Data from an additional 300 non-depressed subjects will be used from ADNI studies for comparison.

Depression history, symptom severity and health information will be collected at the initial visit to determine eligibility. An magnetic resonance imaging (MRI) scan, as well as amyloid (florbetapir) and tau (flortaucipr) positron emission tomography (PET) imaging will be conducted at San Francisco VA. Collection of plasma and serum for biomarkers, clinical assessments and cognitive assessments will be conducted at two time points. Blood samples will also be collected for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Individual participated in original Characterizing Cognitive Decline in Late Life Depression study or Multimodal MRI Characteristics of Psychotherapy Response in Late Life Depression Study.

Exclusion Exceptions:

1. Antidepressant medication treatment is allowed only if the medication dose is stable for 4 weeks prior to the MRI scan.
2. Psychotherapy interventions is allowed only if they have completed at least 4 weeks of individual or group psychotherapy intervention prior to the MRI scan.
3. Participants taking cognitive enhancing medications will be able to enter the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 120 older adults meeting criteria for Major Depression or Late Life Depression (LLD).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-03-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in neuropsychological measures of executive function as measured by the Digit Symbol Substitution Test using total correct. | 5 years (parent protocol), 5 years (continuation)
  The Digit Symbol subtest is a measure of attention, working memory, and information processing speed. Participants are presented with a stimulus sheet, and asked to write in the correct symbol that corresponds with a number keyed at the top of the page. A scaled score is calculated based on the number of total correct responses.
Rate of Change in expressive language as measured by the Boston Naming Test using total correct. | 5 years (parent protocol), 5 years (continuation)
  Boston Naming Test is a measure of visual confrontation naming requires the subject to name objects depicted in outline drawings. The drawings are graded in difficulty, with the easiest drawings presented first. If a subject encounters difficulty in naming an object, a stimulus cue and/or a phonemic cue is provided. The number of spontaneous correct responses (maximum score = 30) and spontaneous plus semantically-cued correct responses (maximum score = 30) are recorded. The number of perceptual errors, circumlocutions, paraphasic errors, and perseverations can also be used to evaluate the subjects' language performance.
Rate of change in learning and memory as measured by the Rey Auditory Verbal Learning Test using total correct and delayed recall. | 5 years (parent protocol), 5 years (continuation)
  Rey Auditory Verbal Learning Test (AVLT) is a list learning task which assesses multiple cognitive parameters associated with learning and memory. On each of 5 learning trials, 15 unrelated words (all nouns) are presented orally at the rate of one word per second and immediate free recall of the words is elicited. The number of correctly recalled words on each trial is recorded. Following a 20-minute delay filled with unrelated testing, free recall of the original 15 word list is elicited. Finally, a yes/no recognition test is administered which consists of the original 15 words and 15 randomly interspersed distracter words. The number of target "hits" and false positive responses are recorded.
Change in brain structure using magnetic resonance imaging (MRI) | 5 years (parent protocol), 5 years (continuation)
  MRI will be used to conduct cortical thickness analysis of whole brain and hippocampus utilizing the following sequences: 3D T1-weighted volume, FLAIR, T2*GRE, and Arterial Spin-Labeling (ASL) Perfusion.
Extent of amyloid deposition as measured by florbetapir | 5 years (parent protocol), 5 years (continuation)
  Data from these scans will be collected via standardized uptake value ratios (SUVR) normalized to the cerebellum
Extent of tau deposition as measured by flortaucipr | 5 years (continuation)

SECONDARY OUTCOMES:
Use biomarkers data employed in ADNI-2 and the NIA AD (Alzheimer's Disease) Genetics Consortium to determine the genotypes needed for the genome wide association study (GWAS). | 5 years (parent protocol), 5 years (continuation)
  Data from participants will be entered into the NIH Genome-Wide database and made available to the scientific community.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Mackin, PhD, Study Director — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Lyness JM, Niculescu A, Tu X, Reynolds CF 3rd, Caine ED. The relationship of medical comorbidity and depression in older, primary care patients. Psychosomatics. 2006 Sep-Oct;47(5):435-9. doi: 10.1176/appi.psy.47.5.435. PMID 16959933
- [Background] McCusker J, Cole M, Ciampi A, Latimer E, Windholz S, Belzile E. Major depression in older medical inpatients predicts poor physical and mental health status over 12 months. Gen Hosp Psychiatry. 2007 Jul-Aug;29(4):340-8. doi: 10.1016/j.genhosppsych.2007.03.007. PMID 17591511
- [Background] Gabryelewicz T, Styczynska M, Luczywek E, Barczak A, Pfeffer A, Androsiuk W, Chodakowska-Zebrowska M, Wasiak B, Peplonska B, Barcikowska M. The rate of conversion of mild cognitive impairment to dementia: predictive role of depression. Int J Geriatr Psychiatry. 2007 Jun;22(6):563-7. doi: 10.1002/gps.1716. PMID 17136705
- [Background] Rapp MA, Gerstorf D, Helmchen H, Smith J. Depression predicts mortality in the young old, but not in the oldest old: results from the Berlin Aging Study. Am J Geriatr Psychiatry. 2008 Oct;16(10):844-52. doi: 10.1097/JGP.0b013e31818254eb. PMID 18827231
- [Background] Ganzini L, Smith DM, Fenn DS, Lee MA. Depression and mortality in medically ill older adults. J Am Geriatr Soc. 1997 Mar;45(3):307-12. doi: 10.1111/j.1532-5415.1997.tb00945.x. PMID 9063276
- See also: National Institute of Mental Health — http://www.nimh.nih.gov/
- See also: Laboratory of Neuro Imaging — http://www.loni.usc.edu/
- See also: Alzheimer's Therapeutic Research Institute — http://atri.usc.edu/studies/
- See also: Related Info — https://latelifedepression.ucsf.edu/